CLINICAL TRIAL: NCT04102631
Title: A Prospective, Randomized, Single-blind, Parallel-controlled Multicenter Study Evaluating the Effectiveness of Endo.Angel in Improving the Quality of Colonoscopy
Brief Title: A Multicenter Study Evaluating the Effectiveness of Endo.Angel in Improving the Quality of Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yu Honggang, Chief of Department of Gastroenterology, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EA-18-002
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Adenoma Detection Rate
Keywords: colonoscopy; computer vision; adenoma detection rate; Endo.Angel
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exposed group (Experimental): patients will receive colonoscopy with assistance of Endo.Angel
  Interventions: Diagnostic Test: colonoscopy with assistance of Endo.Angel
- non-exposed group (Sham Comparator): patients will receive colonoscopy without assistance of Endo.Angel
  Interventions: Diagnostic Test: colonoscopy without assistance of Endo.Angel

INTERVENTIONS:
Diagnostic Test: colonoscopy with assistance of Endo.Angel — Patients in exposed group will receive colonoscopy with assistance of Endo.Angel,a real-time quality monitoring system based on computer vision,which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.
  Arms: exposed group
Diagnostic Test: colonoscopy without assistance of Endo.Angel — Patients in non-exposed group will receive colonoscopy without assistance of Endo.Angel.
  Arms: non-exposed group

SUMMARY:
Colonoscopy is a key technique in the detection and diagnosis of lower gastrointestinal diseases. High quality endoscopy results in better disease outcomes. However, the operant level of different endoscopists is significantly different.This study aims to construct a real-time quality monitoring system based on computer vision, named Endo.Angel, which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.

DETAILED DESCRIPTION:
This study aims to construct a real-time quality monitoring system based on computer vision, named Endo.Angel, which is used to monitor the velocity of insertion of the endoscope, record the time of insertion and withdrawal of the endoscope, and remind endoscopists of the blind areas caused by intestinal segment slipping.Criteria for inclusion and exclusion are determined prior to endoscopic examination. Candidates who meet all inclusion criteria as well as do not meet all exclusion criteria are bring into the study. Participants randomized before the examination, they are divided into the exposed group assisted by Endo.Angel or the non-exposed group without Endo.Angel. Followup are conducted after the examination.Study will be finished when all followup is done,and the examination result collected from participants will send to an independent review data analysis group.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 18 years or above;
2. Colonoscopy is needed to further characterize gastrointestinal diseases;
3. Ability to read, understand and sign informed consent forms;
4. The researchers believe that the subjects can understand the process of the clinical study and are willing and able to complete all the study procedures and follow-up visits to cooperate with the study procedures.

Exclusion criteria:

1. Participated in other clinical trials, signed informed consent forms and followed up in other clinical trials.
2. Participate in a drug clinical trial and during the elution period of the trial or control drug
3. Drug or alcohol abuse or mental disorder in the last 5 years;
4. Pregnant or lactating women;
5. Patients with multiple polyp syndrome;
6. Patients with known space-occupying tumor or intestinal stenosis;
7. Patients with known perforation or colonic obstruction;
8. A history of anaphylaxis with antispasmodic has been documented;
9. The researchers did not consider the subjects suitable for colonoscopy;
10. The researchers determined that the subjects had high-risk diseases or other special conditions that were not appropriate for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1076 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 3 months
  The numerator is the number of cases of adenoma detected by colonoscopy, and the denominator is the total number of cases of patients undergoing colonoscopy.

SECONDARY OUTCOMES:
The mean number of polyps per procedure | 3 months
  The numerator is the total number of polyps detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Polyp Detection Rate | 3 months
  The numerator is the number of patients with polyps detected by colonoscopy, and the denominator is the total number of patients receiving colonoscopy.
The mean number of adenomas per procedure | 3 months
  The numerator is the total number of adenomas detected by colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Detection rate of large, small and minimal polyps | 3 months
  The numerator was the number of patients with large (≥10 mm), small (4-9 mm), and minimal(≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy
The mean number of large, small and minimal polyps per procedure | 3 months
  The numerator was the number of large (≥10 mm), small (4-9 mm), and minimal (≤5 mm) polyps detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of large, small and minimal adenomas | 3 months
  The numerator was the number of patients with large (≥10 mm), small (4-9 mm), and minimal(≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy
The mean number of large, small and minimal adenomas per procedure | 3 months
  The numerator was the number of large (≥10 mm), small (4-9 mm), and minimal (≤5 mm) adenomas detected by colonoscopy, and the denominator was the total number of patients receiving colonoscopy.
Detection rate of adenoma in different sites | 3 months
  The numerator is the number of cases of adenoma detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
The mean number of adenomas in different sites per procedure | 3 months
  The numerator is the total number of adenomas detected in the rectum, sigmoid colon, descending colon, transverse colon, ascending colon and ileocecal region during colonoscopy, and the denominator is the total number of patients undergoing colonoscopy.
Time of colonoscopic withdrawal | 3 months
  the duration of colonoscopic withdrawal(not include the time of biopsy or treatment).
Time of colonoscopic insertion | 3 months
  The time of colonoscopy from the rectum to the ileocecal area.
The rate of reaching the ileocecal region | 3 months
  The numerator is the number of cases of colonic examination reaching the ileocecal region, and the denominator is the total number of colonoscopy cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China